CLINICAL TRIAL: NCT05305118
Title: Safety, Feasibility, and Efficacy of Transcutaneous Spinal Cord Stimulation on Stabilizing Blood Pressure for Acute Inpatients With Spinal Cord Injury
Brief Title: TSCS for Acute SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jill Wecht, Professor, Rehabilitation Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-21-01475; 1648740 (Other: James J. VA Medical Center)
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Acute Spinal Cord Injury; Blood Pressure; Hypotension
Keywords: Transcutaneous Spinal Cord Stimulation; Neuromodulation; Spinal Cord Stimulation; Blood Pressure Disorders; Cerebral Blood Flow Velocity; Acute Inpatient Rehabilitation
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Acute Inpatients With Spinal Cord Injury (Experimental): Inpatient participants undergoing rehabilitation after acute traumatic SCI.
  Interventions: Procedure: TSCS Mapping; Device: Transcutaneous spinal cord stimulation

INTERVENTIONS:
Procedure: TSCS Mapping — Prior to TSCS Intervention, participants will undergo TSCS Mapping.
  Electrode location, pulse frequency will be maintained while the stimulation intensity is ramped from 10 to 200 mA. Brachial blood pressures and symptoms will be monitored and recorded at each ramping interval and will continuously monitor and record beat-to-beat heart rate and blood pressures to determine the optimal site and frequency for further TSCS intervention
  TSCS electrodes will be placed at two vertebral levels in the and back and pulse frequency will be set at 30 to 240 Hz to determine the optimal site and frequency for further TSCS intervention.
Device: Transcutaneous spinal cord stimulation — TSCS will be used as an adjunct intervention to promote blood pressure stability in conjunction with daily physical and occupational therapy in the inpatient rehabilitation gym. Stimulation will be added to therapy 3-5 times per week as needed for the duration of inpatient hospitalization following SCI.
  TSCS stimulation will be delivered using Digitimer DS7A, DS8R stimulators and Chattanooga Continuum (DS7A has FDA 510(k) clearance #K051357; Chattanooga Continuum is a Class 2 device).
  Other Names: TSCS

SUMMARY:
This project will focus on a novel approach to stabilizing blood pressure (BP) during inpatient rehabilitation after acute SCI. After SCI, people have unstable blood pressure, ranging from too low (orthostatic hypotension) to too high (autonomic dysreflexia). Unstable BP often interferes with performing effective physical rehabilitation after SCI. A critical need exists for the identification of safe, practical and effective treatment options that stabilize BP after traumatic SCI. Transcutaneous Spinal Cord Stimulation (TSCS) has several advantages over pharmacological approaches: (1) does not exacerbate polypharmacy, (2) can be activated/deactivated rapidly, and (3) can be applied in synergy with physical exercise. The study team is asking the key question: "What if applying TSCS earlier after injury could prevent the development of BP instability?" To facilitate adoption of TSCS for widespread clinical use, the study team plans to map and develop a parameter configuration that will result in an easy to follow algorithm to maximize individual benefits, while minimizing the burden on healthcare professionals. This project will provide the foundational evidence to support the feasible and safe application of TSCS in the newly injured population, thereby overcoming barriers to engagement in prescribed inpatient rehabilitation regimens that are imposed by BP instability.

DETAILED DESCRIPTION:
This site-specific project will focus on a novel non-pharmacologic approach to stabilizing blood pressure (BP) during acute inpatient rehabilitation after acute traumatic spinal cord injury (SCI). Current forms of pharmacologic and non-pharmacologic treatments for hypotension and orthostatic hypotension remain inadequate in the SCI population. A critical need exists for the identification of safe, practical and effective treatment options that stabilize BP after traumatic SCI as low BP limits the ability of individuals from fully participating in acute rehabilitation therapies. Transcutaneous Spinal Cord Stimulation (TSCS) has several advantages including being able to be activated/deactivated rapidly and the ability to be used during inpatient therapy for rehabilitation following SCI. The study team is asking the key question: "What is the safety and feasibility of applying TSCS in acute SCI to prevent the development of BP instability?" To facilitate adoption of TSCS for widespread clinical use, the study team has designed a mapping and parameter configuration protocol to develop a standard, easy to follow algorithm that will maximize individual benefits of spinal neuromodulation, while minimizing the burden on healthcare professionals. This project will provide the foundational evidence to support the feasible and safe application of TSCS in the newly injured SCI population, thereby overcoming one of the major barriers (i.e., low BP) that prevents full participation in acute SCI rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* All newly injured patients with SCI who are sequentially admitted during the 42-month recruitment period
* Meet the following Model Systems entry criteria with evidence of BP instability
* Exhibit one or more of the following: Resting hypotension - systolic BP ≤ 110 mmHg for males or ≤ 100 mmHg for females; OH - fall in systolic BP ≥ 20 mmHg and/or a fall in diastolic BP ≥ 10 mmHg within 10 minutes of assuming an upright position; BP instability - fluctuation in systolic BP ≥ 20 mmHg and/or fluctuation in diastolic BP ≥ 10 mmHg within a single day during routine activities in the AIR setting.
* Have trouble with your blood pressure as determined by your doctor.
* Participants must be between the ages of 18-89 years old, experienced a spinal cord injury (SCI) within the past 30 days to 6 months, have sustained a SCI with temporary or permanent loss of sensory and/or motor function, and are an inpatient for acute SCI rehabilitation therapy at Mount Sinai.
* You are not dependent on a ventilator at this time.
* You do not have a history of implanted pacemaker/defibrillator or significant coronary artery disease.

Exclusion Criteria:

* Implanted brain/spine/nerve stimulators, cochlear implants, cardiac pacemaker/defibrillator, or intracardiac lines
* Open skin lesions on or near the electrode placement sites (neck, upper back)
* Significant coronary artery or cardiac conduction disease
* Recent history of myocardial infarction
* Insufficient mental capacity to understand and independently provide consent
* Pregnancy
* Cancer
* Deemed unsuitable by study physician

As part of the feasibility assessment, the study team will document demographic and injury characteristics of eligible patients who refuse enrollment, as well as reasons for ineligibility among those who do not meet entrance criteria.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Sit-up Test - Blood Pressure (BP) with and without stimulation. | weekly until discharge, average of 3 weeks
  A brachial BP cuff (Series 400, GE Healthcare, Milwaukee, WI, USA) a finger BP monitor (Finometer ® MIDI Model-2; Finopres Medical Systems BV, Amsterdam, The Netherlands) will be applied. Brachial BP will be monitored at 1-minute intervals for 10-minutes in the supine and 10-minutes in the seated positions.
Severity of Dizziness Scale | weekly until discharge, average of 3 weeks
  The severity of orthostatic dizziness will be assessed at 0, 3, 7 and 10 minutes during the seated BP assessment using a scale from 0 to 10, where 0=no dizziness and 10=severe dizziness.
Sit-up Test - Heart Rate (HR) with and without stimulation. | weekly until discharge, average of 3 weeks
  A 3-lead electrocardiogram (ECG) (RESP1 Impedance Pneumograph, Moro Bay, CA, USA) will be used to determine HR and to estimate parameters of autonomic cardiac control with the recording electrode in the V5 position (immediately below the left anterior axillary line on the same horizontal plane as the 5th intercostal space).

SECONDARY OUTCOMES:
Pain Numeric Rating Scale (NPRS) | weekly until discharge, average of 3 weeks
  Pain scale from 0-10, with higher score indicating more severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Jill Wecht, EdD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Spinal Cord Injury Model System, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. To achieve aims in the approved proposal. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link to be tbd).